CLINICAL TRIAL: NCT00368719
Title: APPLES: A Prospective Pediatric Longitudinal Evaluation To Assess The Long Term Safety Of Tacrolimus Ointment For The Treatment Of Atopic Dermatitis
Brief Title: Evaluation to Assess the Long Term Safety of Tacrolimus Ointment for Atopic Dermatitis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: withdrawn due to contractual issues
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 200614402-1
Record Dates: First submitted 2006-08-24; First posted 2006-08-25 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Tacrolimus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (No Intervention)
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Participants will be followed for 10 years to study the effects of Tacrolimus.

SUMMARY:
To assess the long-term safety of tacrolimus ointment

DETAILED DESCRIPTION:
To assess the long-term safety of tacrolimus ointment 0.03% or 0.1% in the treatment of subjects with atopic dermatitis under actual use conditions, including the risk of developing cutaneous or systemic malignancies. The FDA and EMEA approved Tacrolimus ointment, 0.03% in children and 0.1% and 0.03% in adults, for the treatment of atopic dermatitis. As part of the approval process, the FDA and EMEA requested a post-marketing commitment regarding the safety of long-term use of Tacrolimus ointment in pediatric atopic dermatitis subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject has/had atopic dermatitis.
* Subject has applied tacrolimus ointment 0.03% or 0.1% for at least 6 weeks, continuously or intermittently. This may include subjects who have been enrolled in previous tacrolimus ointment studies and/or subjects with commercial product exposure prior to study enrollment.
* Subject age at the first tacrolimus ointment exposure is/was <16 years of age.
* Subject/Caregiver has given written informed consent and assent as required by state and/or governmental laws, including access to all relevant clinical and medication data, and the storage and analysis of these data.
* Subject/Caregiver agrees to comply with the program requirements including an annual physical exam and biennial dermatological exam and agrees to be contacted and provide information as described in this document to Primary Investigator Dr. Lamb and Covance Periapproval Services, Inc.

Exclusion Criteria:

* Subjects who do not have/ have not had Atopic Dermatitis.
* Subjects must have used Tacrolimus ointment prior to age 16.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2007-09; Study Completion 2016-07

PRIMARY OUTCOMES:
The purpose of this study is to identify the long term effects of Tacrolimus in pediatric subjects | 10 Years

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Tong Liu, M.D., Ph.D., Principal Investigator — Physician with UC Davis Department of Dermatology

REFERENCES:
- See also: University of California-Davis Department of Dermatology Clinical Research — http://www.ucdmc.ucdavis.edu/dermatology/research/clinical